CLINICAL TRIAL: NCT06075784
Title: The Effect of Reiki on Pain, Stress and Comfort Level in Students Experiencing Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Ph.D., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/9
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Therapeutic Touch; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki (Experimental): The intervention will be applied to the reiki group to be applied in the application laboratory of the midwifery department of the faculty of health sciences. Reiki therapy will be applied by a practitioner with a Reiki application certificate in the application laboratory for 30 minutes while the participants lie down with their eyes closed. 4 sessions of reiki application will be applied to the intervention group for a month. Reiki application will start from the time of menstruation, the first pain scores and comfort conditions will be recorded. Menstruation and general comfort after 4 sessions will be recorded. Any medication and side effects during menstruation with the last reiki application will be recorded by the research team member.
  Interventions: Other: reiki
- Placebo reiki (Placebo Comparator): Placebo Reiki will be applied to the participants in the group in the application laboratory of the midwifery department of the faculty of health sciences. The practice will be carried out in the application laboratory for 30 minutes, with the participants sitting with their eyes closed. Reiki life energy will not be transferred to participants in the placebo reiki group. Since the participants' eyes are closed, they will not know that there is a transfer. Placebo Reiki application will be performed in the laboratory 4 times during a month. Placebo application will start from the time of menstruation, and the first pain scores and comfort conditions will be recorded. After 4 sessions, menstruation and general comfort will be recorded. Any medication and side effects during menstruation with the last application will be recorded by the research team member.
  Interventions: Other: reiki

INTERVENTIONS:
Other: reiki — placebo reiki
  Other Names: control group

SUMMARY:
The aim of this study is to determine the effect of reiki on pain, stress and comfort level in students experiencing dysmenorrhea

DETAILED DESCRIPTION:
Hypotheses 01; there was no difference between the pain score of the reiki group and the pain score of the control group.

H02; there was no difference between the stress score of the reiki group and the stress score of the control group.

H03;there was no difference between the comfort level of the reiki group and the comfort level of the control group.

The study will be carried out in two different groups. The practice will start with meeting the students who experienced dysmenorrhea. After the women are evaluated in terms of eligibility criteria for the research, the women who are eligible will be informed about the research and written informed consent will be obtained from the women who accept. The random distribution of women to the study groups will be carried out using the Block Randomization method. The following applications will be made to the groups.

Reiki Group The intervention will be applied to the reiki group to be applied in the midwifery department application laboratory. Reiki therapy will be applied by a practitioner with a Reiki application certificate in the application laboratory for 30 minutes while the participants lie down with their eyes closed. 4 sessions of reiki application will be applied to the intervention group for a month. Reiki application will start from the time of menstruation, the first pain scores and comfort conditions will be recorded. Menstruation and general comfort after 4 sessions will be recorded. Any medication and side effects during menstruation with the last reiki application will be recorded by the research team member.

Placebo Reiki will be applied to the participants in the group in the application laboratory of the midwifery department of the faculty of health sciences. The practice will be carried out in the application laboratory for 30 minutes, with the participants sitting with their eyes closed. Reiki life energy will not be transferred to participants in the placebo reiki group. Since the participants' eyes are closed, they will not know that there is a transfer. Placebo Reiki application will be performed in the laboratory 4 times during a month. Placebo application will start from the time of menstruation, and the first pain scores and comfort conditions will be recorded. After 4 sessions, menstruation and general comfort will be recorded. Any medication and side effects during menstruation with the last application will be recorded by the research team member.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research and volunteering,
* over 18 years of age,
* without a diagnosed psychiatric disease,
* without communication problems,

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Dysmenorrhea
Enrollment: 60 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in pain | immediately before reiki application and immediately after the reiki application
  The Visual Analog Scale is a unidimensional scale commonly used to measure pain intensity. VAS is a measuring tool with a length of 0-10 cm (0-100 mm). This measuring tool can be used horizontally or vertically. High scores from the scale indicate high pain intensity. The cut-off points for pain scores taken from the scale are recommended as 0-4 mm "no pain", 5-44 mm "mild pain", 45-74 mm "moderate pain" and 75-100 mm "severe pain"VAS is a 10-cm-long measurement tool. The left end of the scale reads "no pain at all" and the right end reads "the most intense pian possible". A high score on the scale indicated a high level of pain and a score of 0 pointed to no pain.
Change in stress | immediately before reiki application and immediately after the reiki application
  The Perceived Stress Scale (PSS-10), developed by Cohen, Kamarck and Mermelstein (1983), consists of 14 items in its original form. A self-report style is the scale. The extent to which an individual perceives some situations in his or her life as stressful It measures. For each item, "Never (0)", "Almost never (1)", "Sometimes" 5-point Likert type scoring ranging from "(2)", "Quite often (3)" and "Very often (4)" It is evaluated based on . In the scale, "perception of inadequacy" and "perception of stress/discomfort"
  There are two different factors:
Change in Comfort Level | immediately before reiki application and immediately after the reiki application
  The scale, which was developed by Katharine Kolcaba in 1992 to determine the comfort needs of individuals and to evaluate nursing interventions that can provide comfort and the increase in comfort, was adapted to Turkish society by Kuğuoğlu and Karabacak in 2004. The scale, which is a four-point Likert type and consists of 48 items, was created by taking as a guide the taxonomic structure consisting of 3 levels and 4 dimensions consisting of the theoretical components of comfort. Level; While it is evaluated as relief (16 items), relaxation (17 items) and overcoming problems (15 items), the dimension is; It is evaluated in three parts: physical (12 items), psychospiritual (13 items) and socio-cultural (10 items). Negative expressions in the scale are calculated by reverse coding during the evaluation phase. While the lowest total score that can be obtained from the scale is 48, the highest total score is 192.

CONTACTS AND LOCATIONS:
Overall Officials: Serap TOPATAN, assoc. prof. dr, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)